CLINICAL TRIAL: NCT06203938
Title: Social and Behavioral Associations With Prefrontal Photobiomodulation in Autism Spectrum
Brief Title: Autism Research Project With Non-Invasive Near-Infrared Light Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Francisco Gonzalez-Lima, PhD, Professor, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00005301
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The investigators propose to study the effects of non-invasive transcranial infrared light stimulation (TILS) on individuals with ASD using cognitive testing, questionnaires, and non-invasive near-infrared spectroscopy (NIRS). Participants will have the brain activity monitored by NIRS before and after TILS. Cognitive testing and questionnaires before and after TILS will measure beneficial effects of TILS on cognition and ASD symptoms. TILS will be administered with light-emitting diodes (LEDs), which have general FDA clearance as safe for use in humans.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TILS-treated (Experimental): Transcranial infrared light stimulation (TILS) will be administered via light-emitting diodes (LEDs), which are a safe and non-invasive form of transcranial photobiomodulation.
  Interventions: Device: Transcranial infrared light stimulation
- Sham (Sham Comparator): The sham control group undergoes the same procedure as the treatment group, but without the LEDs turned on.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcranial infrared light stimulation — Trancranial infrared light stimulation administered via light-emitting diodes
  Arms: TILS-treated
Device: Sham — Identical to TILS, but with lights off
  Arms: Sham

SUMMARY:
The investigators have previously shown that the administration of low-level infrared light is a safe and non-invasive procedure which improves cognition and emotion, as well as enhances brain metabolic activity. Based on previous studies, the investigators hypothesize that this methodology, called low-level light therapy or photobiomodulation, could be used to improve behavioral symptoms in individuals with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
The Gonzalez-Lima Laboratory at the University of Texas at Austin will be recruiting participants for a study investigating whether transcranial infrared light stimulation, or TILS, is beneficial for people diagnosed with autism spectrum disorder (ASD).

The molecular target of TILS is cytochrome c oxidase, a mitochondrial enzyme which is crucial for oxygen utilization. People with ASD show impaired mitochondrial function (Siddiqui, Elwell, and Johnson, 2016), as well as alterations in the prefrontal cortex (Amaral, Schumann, and Nordahl, 2008), which plays a key neurological role in mediating attention, impulse control, and social cognition functions.

The lab has previously shown that TILS, delivered to the prefrontal cortex, can be used to improve cognitive functions such as attention (Barrett and Gonzalez-Lima, 2013), executive function (Blanco, Maddox, and Gonzalez-Lima, 2017), and emotional regulation (Zaizar, Papini, Gonzalez-Lima, and Telch, 2021). This cognitive enhancement from TILS is accompanied by an increase in oxygenation of the prefrontal cortex (Holmes, Barrett, Saucedo, O'Connor, Liu, and Gonzalez-Lima, 2019). Recently, the beneficial effects of TILS on ASD symptoms have been safely explored in adults (Ceranoglu et al., 2022) and children/adolescents (Pallanti et al., 2022).

The goal of the study is to recruit children, adolescents, and adults, either ASD or non-ASD, for a study of the effects of repeated administration of TILS on autistic behavior. Participants will be asked to give informed consent, complete a series of questionnaires and cognitive tests, and wear a headband to non-invasively monitor brain activity using near-infrared spectroscopy. TILS is administered non-invasively with a headband device that uses light-emitting diodes (LEDs), which are cleared as safe for use in humans by the Food and Drug Administration (FDA), but the device has not been approved by the FDA for the specific investigational use in this research. The study will train participants (or caregivers) on how to use the LED device, then send the participants home to use the LED device. The investigators will contact participants once a week to check progress. At the end of the study, participants return for the same assessments, at which time the participants will return the LED device.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4-60 years

Exclusion Criteria:

* Current pregnancy

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Autism spectrum questionnaires | Up to two months
  Assess individual differences and changes in autistic traits

SECONDARY OUTCOMES:
Functional near-infrared spectroscopy | Up to two months
  Brain resting state and activational state measures
Continuous Performance Task | Up to two months
  Measure of inattention, impulsivity, sustained attention, vigilance

CONTACTS AND LOCATIONS:
Overall Officials: Sarah W Diaz, PhD, Study Director — University of Texas at Austin
Locations (1):
- Seay Psychology Building, Room 3.304, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
What data will be shared? Individual participant data that underlie the results reported in this study, after deidentification (text, tables, figures, and appendices).
  A data dictionary, including a description of the variables and types of data, collected for each individual, will be provided. This data will include anonymized individual participant demographic information and all outcome variables (cognitive task data, spectroscopy data).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The raw data will be made available by the researchers upon reasonable request by any qualified doctoral researcher (PhD, MD). They will be granted access by contacting the corresponding author/principal investigator (F. Gonzalez-Lima, utbrainproject@gmail.com).
  It will be made available to qualified researchers whose proposed use of the data has been approved by an independent review committee (Institutional Review Board) identified for the purpose of individual participant data meta-analysis.
  Proposals may be submitted up to 36 months following article publication. After 36 months, the data will be available in our University's shared network drive, but without investigator support other than deposited metadata.
URL: https://labs.la.utexas.edu/gonzalez-lima/idp-plan/